CLINICAL TRIAL: NCT02183350
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses (1, 2.5, 5, 10 and 25 mg q.d. for 12 Days) of BI 1356 BS as Powder in the Bottle (PIB) in Patients With Type 2 Diabetes (Randomised, Double-blind, Placebo-controlled Within the Dose Groups).
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 1356 BS in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.2
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- BI 1356 BS - single rising dose (Experimental)
  Interventions: Drug: BI 1356 BS - single rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1356 BS - single rising dose
  Arms: BI 1356 BS - single rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the current study was to investigate the safety and tolerability of BI 1356 BS following administration of multiple rising oral doses of 1 mg, 2.5 mg, 5 mg, and 10 mg over 12 days in male patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Male patients with proven diagnose of type 2 diabetes mellitus treated with diet and exercise only or with one (or two) oral hypoglycaemic agents besides glitazones

* Glycosylated haemoglobin A1 (HbA1c)

  * ≤ 8.5 % at screening for patients treated with diet and exercise and/or one oral hypoglycaemic agent or
  * ≤ 8.0 % at screening for patients treated with two oral hypoglycaemic agents
* Age ≥21 and Age ≤65 years
* BMI ≥18.5 and BMI ≤35 kg/m2 (Body Mass Index)
* Caucasian ethnicity
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice GCP and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including Blood Pressure (BP), Pulse Rate (PR) and Electrocardiogram (ECG)) deviating from normal and of not acceptable clinical relevance
* Clinically relevant concomitant diseases like renal insufficiency, cardiac insufficiency New York Heart Association (NYHA) II-IV, known cardiovascular diseases including hypertension > 160/110 mmHg, stroke and Transient ischaemic attack (TIA)
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders besides type 2 diabetes, hyperlipidaemia and medically treated hypertension
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or relevant neurological disorders besides polyneuropathy
* Chronic or relevant acute infections (e.g. Human immunodeficiency virus (HIV), Hepatitis)
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial except allowed co-medication
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of not acceptable clinical relevance
* Change of drug dosing of allowed co-medication (anti-hypertensive agents, acetylic salicylic acid and statins) within the last 3 months
* Any ECG value outside of the reference range and of clinical relevance including, but not limited to QRS interval > 120 ms or QTcB > 450 ms or QT >500 ms
* Fasted blood glucose > 240 mg/dl (=13.3 mmol/L) on two consecutive days during washout
* Serum creatinine above upper limit of normal at screening

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-04; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 28 days
Number of patients with abnormal findings in physical examination | up to 28 days
Number of patients with abnormal changes in Vital signs (blood pressure (BP), pulse rate (PR)) | up to 28 days
Number of patients with abnormal changes in 12-lead ECG (electrocardiogram) | up to 28 days
Number of patients with abnormal changes in laboratory parameters | up to 28 days
Assessment of tolerability by investigator on a 4-point scale | up to 28 days

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | predose, up to 456 h
tmax (time from dosing to maximum concentration) | predose, up to 456 h
AUC (area under the concentration-time curve of the analyte in plasma) | predose, up to 456 h
Ae (amount of analyte that is eliminated in urine) | predose, up to 456 h
fe (fraction of analyte excreted in urine) | up to 288 h
CLR (renal clearance of the analyte in plasma) | up to 288 h
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval) | predose, up to 456 h
Cpre,N (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose N) | predose, up to 456 h
λz,ss (terminal rate constant in plasma at steady state) | predose, up to 456 h
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | predose, up to 456 h
MRTpo,ss (mean residence time of the analyte in the body after 12 administrations at steady state) | predose, up to 456 h
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | predose, up to 456 h
Vz/F,ss (apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state) | predose, up to 456 h
Changes in PTF (peak trough fluctuation) | up to 28 days
RA,Cmax based on Cmax | predose, up to 456 h
RA,AUC based on AUCτ | predose, up to 456 h
Changes in Dipeptidyl-Peptidase IV (DPP-IV) activity in plasma | predose, up to 456 h
Change in plasma glucose levels | up to 13 days